CLINICAL TRIAL: NCT05067582
Title: A Randomized, Double-Blind, Chronic Dosing (12-weeks), Two-Period, Placebo-Controlled, Crossover, Multi-Center Study to Assess the Efficacy, Safety, and Tolerability of Two Doses of L1-79 for the Treatment of the Core Deficits in Social-Communication Interaction in Adolescents and Young Adults With Autism Spectrum Disorder
Brief Title: A 12-Week Crossover Study to Assess the Efficacy, Safety and Tolerability of L1-79 in Subjects Aged 12-21 Years With Autism Spectrum Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yamo Pharmaceuticals LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Y202
Record Dates: First submitted 2021-09-22; First posted 2021-10-05 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Autism Spectrum Disorder; Autism
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Intervention Model Description: Two Period Crossover
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo Capsules (Placebo Comparator): 1 capsule twice daily
  Interventions: Drug: L1-79
- L1-79 200 mg or 300 mg Capsules (Experimental): 1 capsule twice daily
  Interventions: Drug: L1-79

INTERVENTIONS:
Drug: L1-79 — tyrosine hydroxylase inhibitor
  Other Names: DL-alpha-Methyltyrosine

SUMMARY:
This study will investigate the efficacy, safety and tolerability of L1-79 in participants aged 12-21 years who have been diagnosed with ASD with a score of >/= 70 on the Wechsler Abbreviated Scale of Intelligence (WASI-II), and a score of >/= 4 on the Clinical Global Impression of Severity of Illness (CGI-S) weighted for socialization.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adolescents or young adults between 12 and 21 years of age.
* WASI-II standard score with 95% CI containing 70 or greater at screening or within the last 12 months prior to screening.
* Fulfill language criteria required to complete ADOS-2 Modules 2, 3 or 4.
* Diagnosis of ASD based on tool that utilizes the DSM-5 criteria, confirmed with ADOS-2.
* CGI-S (weighted for socialization) of 4 or greater.
* A female is eligible to enter and participate in the study if she is of non-childbearing potential or childbearing potential, has negative pregnancy test at screening and, if sexually active, agrees to use acceptable contraception methods (defined in protocol), for the duration of the study and for at least 30 days after the last dose of study drug.
* Male subjects if sexually active and female partners of childbearing potential must agree to use acceptable contraceptive methods (defined in protocol), for the duration of the study and for at least 30 days after the last dose of study drug.
* Subjects and caregiver must be willing and able to participate in the testing procedures sufficient to obtain valid scores on the tests used herein.
* Must live with a parent/primary caregiver, or if not, during each week he/she must either spend at least 3 hours a day for at least 4 days or, spend the weekend with a parent/primary caregiver.
* In the opinion of the Investigator, be sufficiently tolerant and capable of complying with the requirements of this trial.
* Able to swallow study medication whole and self-administer medication if living independently or have a parent/caregiver be able to administer medication.
* Subjects or their legal guardians must be willing to sign informed consent and/or assent and caregivers participating in the study must be willing to sign informed consent.

Exclusion Criteria:

* Pregnancy or breastfeeding, or intention to become pregnant during the study.
* Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic cardio-vascular disease, hepatic disease, renal disease, musculo skeletal or rheumatologic disease, human immunodeficiency virus (HIV), hemorrhagic cerebrovascular accident (HCVA), hepatitis B virus (HBV), or psychiatric illness/social situations that would limit compliance with study requirements.
* Any disease that requires treatment with immunosuppressive drugs.
* A diagnosis of Fragile-X syndrome or Rett syndrome.
* A DSM-5 diagnosis of schizophrenia, schizoaffective disorder, alcohol use disorder, current or lifetime diagnosis of severe psychiatric disorder (e.g., bipolar disorder, etc.).
* Subjects at risk of suicidal behavior or with a history alcohol or substance abuse/dependence.
* Presence of any active chronic medical problem including, but not limited to uncontrolled: seizure disorder, heart disease, cancer, asthma, genetic disease.
* Requiring more than 3 medications for the treatment of autism, ADHD, seizures, depression, anxiety, aggression, agitation, obsessive compulsive disorder, tic disorder, or other disorder commonly co-occurring with ASD.
* Initiation of new or major change in psychosocial intervention within 12 weeks prior to screening and throughout the duration of the study.
* School or academic setting are expected to change during the course the study.
* Clinically significant ECG abnormalities including subjects with baseline QTc prolongation (QTcF >450 msec for males and >470 msec in females).
* On concomitant medications known to prolong the QTc interval.
* Presence of out of range hepatic or renal function tests or other unexplained abnormal laboratory value that is deemed clinically significant by the Investigator.
* On any of the following medications: alpha-2 agonists (including, but not limited to clonidine and guanfacine), beta-blockers, anti-hypertensives, and antipsychotics not approved for use in ASD.
* Taking disallowed concomitant medications within 2 months (antipsychotics) and 1 month (all other medications) prior to Baseline.
* Any subject or caregiver who is unwilling or unable to give informed consent.
* Participated in an investigational drug study within 90 days prior to Baseline.

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 58 (Actual)
Dates: Start 2022-01-25 (Actual); Primary Completion 2024-06-18 (Actual); Study Completion 2024-06-21 (Actual)

PRIMARY OUTCOMES:
Vineland Adaptive Behavior Scale, Third Edition (Vineland-3), Responder Analysis | Week 12
  at least 1 point improvement in 2/3 socialization subdomains or at least 3 point improvement in socialization domain

SECONDARY OUTCOMES:
Vineland-3 Socialization Domain, Standard Score | Week 12
V-scale Score for Each of the 3 Socialization Subdomains of the Vineland-3 | Week 12
Clinical Global Impression of Severity of Illness (CGI-S) Weighted for Socialization | Week 12
Clinical Global Impression of Change (CGI-C) Weighted for Socialization | Week 12
Growth Scale Value (GSV) of Each of the 3 Socialization Subdomains of the Vineland-3 | Week 12
Caregiver Global Impression of Change of 3 Most Bothersome Symptoms of ASD (CGI-3P) | Week 12
Social Responsiveness Scale, Second Edition (SRS-2) Social-Communication and Interaction - DSM-5 Composite T-score | Week 12
Social Responsiveness Scale, Second Edition (SRS-2) Social Awareness T-score | Week 12
Social Responsiveness Scale, Second Edition (SRS-2) Social Cognition T-score | Week 12
Social Responsiveness Scale, Second Edition (SRS-2) Social Motivation T-score | Week 12
Social Responsiveness Scale, Second Edition (SRS-2) Social Communication T-score | Week 12
Social Responsiveness Scale, Second Edition (SRS-2) Total T-score | Week 12
Parent-rated Anxiety Scale for ASD (PRAS-ASD) | Week 12
Aberrant Behavior Checklist, Second Edition (ABC-2) Social Withdrawal/Lethargy Subscale | Week 12
Aberrant Behavior Checklist, Second Edition (ABC-2) Inappropriate Speech Subscale | Week 12
Child's Sleep Habits Questionnaire (CSHQ) | Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Tom Megerian, MD, PhD, Study Director — CMO and Senior VP of Clinical Development
Locations (8):
- United States (8):
  - Southwest Autism Research and Resource Center, Phoenix, Arizona
  - Thompson Autism Center CHOC, Orange, California
  - Cortica, San Rafael, California
  - Rush University, Chicago, Illinois
  - Thompson Center for Autism and Neurodevelopmental Disorders, Columbia, Missouri
  - Center for Autism and The Developing Brain, White Plains, New York
  - Ohio State University, Columbus, Ohio
  - Red Oak Psychiatry Associates, Houston, Texas

IPD SHARING:
Plan to Share IPD: No